CLINICAL TRIAL: NCT06048016
Title: Effect Of Scaling and Root Planning on Alkaline Phosphatase in Saliva and Gingival Crevicular Fluid in Periodontitis Patients Compared With Healthy Subjects Before and After Treatment
Brief Title: Effect Of Scaling and Root Planning on ALP in Saliva and GCF In Periodontitis Patients Compared With Healthy Individuals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Azzahraa Abdel Fattah Abdelrahim, Principle investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PER7_2_1
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Periodontitis; Healthy
Keywords: ALP; Scaling; GCF; Saliva; Periodontitis; Health
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation

STUDY DESIGN:
Intervention Model Description: Group 1 : 68 Periodontitis Patients, providing scaling and root plaining . Group 2:68 healthy individuals.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- periodontitis patients (Experimental): Periodontitis Patients participate to test level of ALP in saliva and GCF.
  Interventions: Diagnostic Test: Scaling and Root Planning

INTERVENTIONS:
Diagnostic Test: Scaling and Root Planning — Scaling and Root Planning by using ultrasonic scaler ,and Gracy currettes.
  Other Names: gingival debridement

SUMMARY:
The goal of this [interventional clinical trial] is to test effect of scaling and root plaining on Alkaline phosphatase in Saliva and Gingival crevicular fluid in periodontitis patients compared with healthy subjects The population from periodontitis patients compared with healthy individuals

It aims to answer are:

• 1_Alkaline phosphatase level in saliva and GCF. 2_Scaling and root plaining effect on Alkaline Phosphatase level. 0 participants will be asked to maintain their oral hygiene instructions.

Researchers will compare [periodontitispatientsto healthyindividuals] to see if [AlkalinePhosphatase level].

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease that destroys the periodontium and is the leading cause of adult tooth loss (Hajishengallis 2014). Periodontitis causes systemic inflammation and immune response via microorganisms and their products in subgingival plaque biofilm, and it is a risk factor for systemic diseases (Lim et al. 2020).

Diagnosis of periodontal disease is made after analyzing the information collected from a periodontal examination. Traditional periodontal diagnostic parameters used clinically include probing depths, bleeding on probing, clinical attachment levels, plaque index and radiographs assessing alveolar bone level (Taba et al. 2005).

The aim of periodontal diagnostic procedures is to provide the clinician with useful information about the current periodontal disease type, location, and severity. These findings form the foundation for treatment planning and provide critical information during the periodontal maintenance and disease-monitoring phases of treatment (Taba et al. 2005).

Traditional diagnostic procedures are inherently limited, in that only disease history, not current disease status, can be assessed. Advances in diagnostic research in oral and periodontal disease are moving toward methods whereby periodontal risk can be identified and quantified by objective measures such as biomarkers (Sanikop S et al.2012).

A biomarker is a substance that indicates a biological state and serves as an objective measure to assess current and future disease activity (Pavankumar et al. 2015). The response of an organism to periodontal infection includes production of several enzymes released from stromal, epithelial, inflammatory, or bacterial cells. These intracellular enzymes are released increasingly from the damaged cells of periodontal tissues into the gingival crevicular fluid (GCF) and saliva (Sanikop S et al.2012).

Saliva contains the body's most important electrolytes (calcium, phosphorous and other minerals). They get a significant impact on the formation, maturation, and metabolism of dental plaque. Salivary calcium and phosphorus concentrations are important for periodontal health because an increased level of salivary calcium or phosphorous is associated with rapidly mineralized plaque, which is associated with poor oral hygiene. As a result, salivary biomarkers such as calcium, phosphorus, alkaline phosphatase, and pH can be used to assess the diagnosis and prognosis of gingivitis or periodontitis(Alaauldeen et a2015).

Gingival crevicular fluid (GCF) has greatly aided our understanding of periodontal disease pathogenesis. A very small amount of fluid analysis may reveal significant clinical changes occurring within the gingiva. These modifications may be useful in the diagnosis of periodontal disease (Koregol et al. 2011). GCF is regarded as a promising medium for the detection of markers of periodontal disease activity. Periodontal diseases are characterised by the destruction of tooth-supporting tissues, and quantitation of tissue breakdown products in GCF has been pursued as a means of identifying active disease sites (Koregol et al. 2011).

Alkaline phosphatase is a catalytic enzyme that accelerates the removal of phosphate groups in the 5 and 3 positions from a wide range of molecules such as nucleotides, proteins, and alkaloids. Although ALP is found in all tissues, it is especially abundant in the bone, liver, bile duct, kidney, and placenta(Pavankumar et al. 2015). It is a membrane bound glycoprotein produced by many cells such as neutrophils during inflammation, osteoblasts during bone production, and periodontal ligament fibroblasts during regeneration. ALP is regarded as a critical indication of osteoblastic activity. The presence of ALP in the saliva and GCF is usually indicative of inflammation and/or destruction of the periodontal tissues. The level of ALP is positively correlated with the severity of the periodontal disease (Pavankumar et al. 2015).

The normal level of ALP in the human blood ranges from 25 to 100 IU/L when the concentration of ALP is higher than 300 IU/L, it is an indicator of several diseases including liver diseases, liver cancer, hepatitis, bone disease, osteoblastic bone cancer (Wang et al., 2009).

ELIGIBILITY:
Inclusion Criteria:

* periodontitis patients stage I,II,III,IV Having more than 10 remaining teeth. • Systemically free

Exclusion Criteria:

* infectious diseases dependent on antibiotics. .inflammatory diseases depend on analgesics. . Diabetes mellites patients . Hypertensive patients

  .Thyroid disease
* Patients who had professional periodontal treatment during the last 6 months.
* Pregnancy or lactation.
* Smokers.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-07-10 (Estimated)

PRIMARY OUTCOMES:
Effect Of Scaling and Root Planning on Alkaline Phosphatase level in saliva and GCF | 1 month
  Measuring ALP level in Saliva and Gingival crevicular before and after treatment

SECONDARY OUTCOMES:
Comparing periodontitis patients to healthy individuals | 1 month
  Compare ALP level in periodontitis patients to healthy individuals

CONTACTS AND LOCATIONS:
Overall Officials: Zahraa Af Nasser, Principal Investigator — Cairo University
Locations (1):
- Zahraa Nasser, Giza, Haram, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The participants data will include their phone numbers,photos, their signature
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 month
Access Criteria: Phone number Consent